CLINICAL TRIAL: NCT04063618
Title: Reduction of Concussion Symptoms Through the Use of Osteopathic Manipulative Therapy: A Prospective Study
Brief Title: Reduction of Concussion Symptoms Through the Use of Osteopathic Manipulative Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient subject enrollment
Sponsor: Matthew T. Mcelroy, DO (Other)
Responsible Party: Sponsor-Investigator, Matthew T. Mcelroy, DO, Staff Physician, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0612
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Therapy (OMT) Treatment Group (Experimental): Initial concussion treatment will involve OMT in addition to standard of care treatment. The OMT practitioner, using a strong anatomic knowledge base, applies specific genital forces in the dysfunctional area, thus providing aid to the body's innate mechanisms of healing. During OMT, a patient's muscles and joints are moved using techniques that include stretching, gentle pressure, and resistance.
  Interventions: Procedure: Osteopathic Manipulative Therapy; Procedure: Standard of Care Concussion Treatment
- Standard of care concussion treatment group (Active Comparator): Standard of care concussion treatment without OMT
  Interventions: Procedure: Standard of Care Concussion Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Therapy — The OMT practitioner, using a strong anatomic knowledge base, applies specific genital forces in the dysfunctional area, thus providing aid to the body's innate mechanisms of healing. During OMT, a patient's muscles, joints, and tissues are moved using techniques that include stretching, gentle pressure, and resistance.
  Arms: Osteopathic Manipulative Therapy (OMT) Treatment Group
Procedure: Standard of Care Concussion Treatment — Standard of care for concussion management is cognitive rest, meaning no stimulation (or as little as possible). This mean no TV/phones/music/school/homework generally for 24 hours. After that a return to academic work is typically started. Once patient is symptom free for 24 hours, then the return to play protocol is initiated (this takes 7 total days to complete at a minimum).

SUMMARY:
Concussion incidence in high school and collegiate sports is high, especially in football. Once diagnosed, return to play is dependent on recovery from symptoms followed by a specific protocol for clearance; the sooner the symptoms subside the sooner the protocol is initiated. Osteopathic Manipulative Therapy (OMT) is a low risk procedure that has minimal side effects and has been used to decrease both headache intensity and frequency. With the main subjective symptom tracked for concussion being headache, OMT may be used to decrease the severity and the duration of this symptom.

DETAILED DESCRIPTION:
Concussion incidence in high school and collegiate sports is high, especially in football. These injuries have become the focus of the sports world, as coaches, trainers, and medical personnel are more vigilant than ever in screening for concussions. Once diagnosed, return to play is dependent on recovery from symptoms followed by a specific protocol for clearance; the sooner the symptoms subside the sooner the protocol is initiated. Osteopathic Manipulative Therapy (OMT) is a low risk procedure that has minimal side effects and has been used to decrease both headache intensity and frequency. With the main subjective symptom tracked for concussion being headache, OMT can be used to decrease the severity and the duration of this symptom. In a prospective superiority comparison between standard of care for concussion (rest and return to play protocol) and a single OMT treatment in combination with standard therapy, we hypothesize that OMT decreases symptom duration and severity of headache in concussion management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to the Geisinger sports medicine clinic or athletic training room for concussion evaluation and management
2. Age less than 25 years old
3. Enrolled in high school or college
4. Participating in a sport at either collegiate or high school level

Exclusion Criteria:

1. Diagnosis does not meet criteria for concussion
2. Symptoms of concussion not present on initial visit
3. Patient unable to tolerate the OMT treatment
4. Patient needs intervention beyond standard concussion management
5. Patients not able to provide consent to be a part of the study

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Concussion Severity Score | 7 days
  Patient will score him or herself on a scale from 0-6 for each of 22 concussion related symptoms. A score of "0" is equal to no symptoms, a score of 1-2 is mild, a score of 3-4 is moderate, a score of 5-6 is severe. Total score is calculated by adding each individual item score. Higher scores are worse than lower scores.
Duration of concussion symptoms | 7 days
  Measured in days; how does Concussion Severity Score change over time
Time to start of the return to play protocol | 7 days
  Measured in days; Once diagnosed, return to play is dependent on recovery from symptoms followed by a specific protocol for clearance; the sooner the symptoms subside the sooner the protocol is initiated.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McElroy, DO, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Woodbine, Danville, Pennsylvania, United States